CLINICAL TRIAL: NCT01659580
Title: Phase III Confirmatory Trial to Confirm the Anti-anginal Effect of Dantonic® (T89) in Patients With Chronic Stable Angina
Brief Title: Phase III Trial of Dantonic® (T89) Capsule to Prevent and Treat Stable Angina
Acronym: CAESA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tasly Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T89-07-CAESA; T89-07-GL (Other: Tasly Pharmaceuticals INC.)
Record Dates: First submitted 2012-07-19; First posted 2012-08-08 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Angina Pectoris
Keywords: Angina Pectoris Treatment Prevention
MeSH Terms: conditions — Angina Pectoris | interventions — T89 herbal drug

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- T89 high dose (Experimental): T89 225mg bid
  Interventions: Drug: T89 high dose
- T89 low dose (Experimental): T89 150mg bid
  Interventions: Drug: T89 Low dose
- Sanqi+Bingpian (Experimental): 225mg bid
  Interventions: Drug: Sanqi+Bingpian
- Placebo (Placebo Comparator): 225mg bid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: T89 high dose — 225mg bid
  Other Names: Dantonic®; Compound Danshen Dripping Pills; Salvtonic®
  Arms: T89 high dose
Drug: T89 Low dose — 150mg bid
  Other Names: Dantonic®; Salvtonic®; Compound Danshen Dripping Pill
  Arms: T89 low dose
Drug: Sanqi+Bingpian — 225 mg bid
  Arms: Sanqi+Bingpian
Drug: Placebo — 225mg bid
  Arms: Placebo

SUMMARY:
This phase III study is designed as a double blind, randomized, multi-nation, multi-center, placebo controlled clinical research, which aims to evaluate the safety and efficacy of Dantonic® (T89) in patients with chronic stable angina pectoris.

DETAILED DESCRIPTION:
Dantonic® (T89) is a botanical drug consists of extracts of Danshen (Radix Salviae Miltiorrhizae) and Sanqi (Radix Notoginseng) with borneol in a capsule form. The drug is currently approved in 26 countries outside the USA for the treatment and prevention of chronic stable angina pectoris and other cardiovascular disease related conditions. This pivotal confirmative Phase III clinical trial is to confirm the efficacy and safety of the drug at 150mg and 225mg doses in the prevention and treatment of angina pectoris in patients with Chronic Stable Angina. The contribution of the main herb Danshen to, and the difference of various production batches in, the overall efficacy and safety profiles will also be explored. Patients will take a morning and an evening dose orally (every 12 hours) for 6 weeks while stop taking any long-acting nitroglycerin, ranolazine, and/or multiple beta-blockers or beta blocker(s) with calcium channel blocker during the trial. Single beta-blocker and/or on-demand short acting nitroglycerin to relief angina pectoris is allowed during the trial. After physical exams and if eligible to participation, patients will stop taking other drugs, and undergo two baseline screen Exercise Treadmill Tests (ETT) on Standard Bruce Protocol in the clinic one week before and right before starting the drug treatment. Patients will perform three more ETTs before the morning dose at the end of week 2, 4 and 6 after receiving the drug treatment. The primary efficiency endpoint is the change of symptom-limited Total Exercise Duration of the ETT at the end of the 4th week of treatment from the average of the two screening baselines compared with that of placebo treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Males and females between the ages of 20 and 80 years.
3. Females of childbearing potential must have a negative pregnancy test, not be breast feeding and established on a method of contraception that in the investigator's opinion is acceptable. Females must agree to remain on their established method of contraception through their participation in the study and for 14 days following the last dose of study drug.
4. Evidence of coronary artery disease that consists of a well-documented medical history (over 3 months prior to the enrolment) of myocardial infarction or significant coronary artery disease with noninvasive or angiographic confirmation.
5. Symptoms that support the diagnosis of chronic angina and/or a history of an abnormal exercise response limited by angina and/or electrocardiograph (ECG) changes.
6. Moderate angina pectoris (Class II or III, Grading of Angina Pectoris by the Canadian Cardiovascular Society Classification System).
7. Patient whose symptom-limited Total Exercise Duration (TED) is between 3 to 7 minutes in Exercise Tolerance Test (ETT) on Standard Bruce Protocol, and symptom-limited TED on two screen examinations (Day -7 and 0) in which the shorter is within 85% of the longer .
8. Patient has been on one beta-blocker or on one calcium-channel blocker for at least 14 days prior to dosing of study medication and can remain on this treatment throughout the study as background anti-anginal treatment. Short-acting nitroglycerin for on-demand use is allowed for all eligible patients.
9. Understand and be willing, able and likely to comply with all study procedures and restrictions and comprehends the verbal rating scales and diary cards.

Exclusion Criteria:

1. With contraindication to, unable to, or with other co-morbidities that may prevent or interfere with the ability to perform treadmill ETT (including, but not limited to: pulmonary hypertension, functionally limiting COPD (chronic obstructive pulmonary disease), history of pulmonary tuberculosis, prior hospitalization for acute exacerbation of chronic lung disease, home oxygen use, chronic oral steroid therapy that can limit exercise capacity, functionally limiting peripheral artery disease, etc.).
2. Presence of electrocardiographic or other abnormalities/factors that could interfere with exercise electrocardiograph interpretation or may lead to a false positive stress test (e.g., pre-exercise horizontal or down-sloping ST segment depression in any standard lead, cardiac glycoside therapy, Lown-Ganong-Levine Syndrome, Wolff-Parkinson-White syndrome (WPW), left bundle branch block, left ventricular hypertrophy with repolarization abnormality, implanted pacemaker, etc.).
3. Clinically significant arrhythmias or atrioventricular conduction block greater than first degree, decompensated heart failure, atrial fibrillation, hypertrophic cardiomyopathy.
4. Acute coronary syndrome (acute myocardial infarction or unstable angina) in the prior 2 months or coronary revascularization within the prior 6 months or planned coronary revascularization during the study period.
5. Congenital cardiac defects, ongoing history of decompensated congestive heart failure, severe valvular disease, severe uncontrolled hypertension (seated systolic blood pressure > 180 mm Hg or diastolic blood pressure > 110 mm Hg), severe anemia, suspected or known dissecting aortic aneurysm, acute myocarditis or pericarditis, thrombophlebitis or pulmonary embolism.
6. History of bleeding diathesis, cerebral hemorrhage, or seizure disorders that required anticonvulsant medication.
7. Patients requiring the use of long-acting nitroglycerin, ranolazine, and/or multiple anti-anginal drugs.
8. Aspirin and/or statins started less than 14 days prior to the signing of informed consent.
9. Pregnancy or lactation.
10. Clinical trials/experimental medication 1) Participation in any other clinical trial or receipt of an investigational drug within 30 days prior to the initial visit.

2) Previous participation in the studies of T89. 11. Substance abuse. Patients with a recent history (within the last 2 years) of alcoholism or known drug dependence.

12. Is a family member or relative of the study site staff. 13. Any other conditions that, in the opinion of the investigator, are likely to prevent compliance with the study protocol or pose a safety concern if the subject participates in the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1004 (Actual)
Dates: Start 2012-08; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The change of symptom-limited TED from baseline compared to placebo at the end of week 4. | 4 weeks
  The change of symptom-limited Total Exercise Duration (TED) at trough drug levels at the end of the 4th week of treatment from screen baseline on Standard Bruce Protocol compared with placebo.

SECONDARY OUTCOMES:
The change of symptom-limited TED at trough drug levels at the end of the 2nd and 6th weeks | 2nd weeks and 6th weeks
  The change of symptom-limited TED at trough drug levels at the end of the 2nd and 6th weeks of treatment from screen baseline on Standard Bruce Protocol compared with placebo;
Frequency of weekly angina episodes | 6 weeks
  Frequency of weekly angina episodes

OTHER OUTCOMES:
Time to onset of angina during Excise Tolerance Test (ETT); | 6 weeks
  Time to onset of angina during ETT;

CONTACTS AND LOCATIONS:
Overall Officials: Henry He Sun, PhD, Study Director — Tasly Group, Co. Ltd.
Locations (94):
- United States (30):
  - Cardiology and Medicine Clinic, Little Rock, Arkansas
  - Beaver Medical Clinic, Banning, California
  - Foundation for Cardiovascular Medicine, La Jolla, California
  - Precision Research Institute, National City, California
  - Paradigm Clinical Research Institute, Inc., Torrance, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Brevard Cardiovascular Research Associates, Merritt, Florida
  - SouthCoast Research Center, Inc, Miami, Florida
  - Molecular Imaging Research and Clinical Trials, Miami, Florida
  - Integrity Clinical Trials, Miami, Florida
  - NewPhase Clinical Trials, Inc., Miami Beach, Florida
  - Peninsula Research, Inc., Ormond Beach, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Jedidiah Clinical Research, Tampa, Florida
  - Athens Heart Center, Athens, Georgia
  - Atlanta Clinical Research Center, Atlanta, Georgia
  - Ellipsis Research, Atlanta, Georgia
  - Central Cardiology, Campbellsville, Kentucky
  - Alexandria Cardiology Clinic, Alexandria, Louisiana
  - Tulane University Health Science Center, Tulane University Heart & Vascular Institute, New Orleans, Louisiana
  - Manhattan Medical Research Practice, New York, New York
  - Cleveland Clinic, Medina, Ohio
  - Hillsboro Cardiology, PC, Hillsboro, Oregon
  - Kore CV Research, Jackson, Tennessee
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - Angiocardiac Care of Texas, PA, Houston, Texas
  - Northwest Houston Cardiology, Houston, Texas
  - Cardiology Center of Houston, PA, Katy, Texas
  - Northwest Heart Center, Tomball, Texas
- Minsk Regional Clinical Hospital, Minsk, Belarus, Belarus
- Canada (14):
  - Dr. Petr Polasek, MD, Office of, Kelowna, British Columbia
  - The Medical Arts Health Research Group, North Vancouver, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - Dixie Medical Group, Mississauga, Ontario
  - Bakbak Medicine Professional Corporation, Oshawa, Ontario
  - Heart Care Research, Oshawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - ViaCar Recherche Clinique Inc., Brossard, Quebec
  - ViaCar Recherche Clinique Inc., Greenfield Park, Quebec
  - Centre Cardiovasculaire De La Rive-Sud (Ccrs), Longueuil, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Clinique Sante Cardio MC, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec, Quebec
  - Centre de Sante et de Services Sociaux de Trois-Rivieres, Trois-Rivières, Quebec
- Georgia (8):
  - The "Unimed Ajara", Batumi, Georgia
  - Cardiological CLinic "Guli" Ltd, Tbilisi, Georgia
  - Archangel St. Michael Multiprofile Clinical Hospital, Tbilisi, Georgia
  - Cardio-Reanimation Centre, Tbilisi, Georgia
  - Emergency Cardiology Center named by Academician G. Chapidze Ltd, Tbilisi, Georgia
  - Tbilis Heart and vascular clinic Ltd., Tbilisi, Georgia
  - Center of Vascular and Heart Diseases Ltd., Tbilisi, Georgia
  - "Clinic L J" Ltd, Tbilisi, Georgia
- Mexico (8):
  - Hospital de Cardiología de Aguascalientes, Aguascalientes, Aguascalientes
  - Centro para el Desarrollo de la Medicina y Asistencia Médica Especializada SC sede Torreon Coahuila, Torreón, Coahuila
  - Consultorio Medico de Especialidad, Tijuana, Estado de Baja California
  - Cardiocen de Guadalajara, S.C., Guadalajara, Jalisco
  - Centro de Investigación Clínica Chapultepec, Morelia, Michoacán
  - OSMO, Oaxaca City, Oaxaca
  - Hospital Central "Dr. Ignacio Morones Prieto", San Luis Potosí City, San Luis Potosí
  - Centro para el Desarollo de la Medicina y de Asistencia Medica Esp. S.C., Culiacán, Sinaloa
- Russia (17):
  - Regional Buegetary Healthcare Institution "Cardiological Dispensary", Ivanovslaya, Ivanovslaya Obl.
  - Nonstate Healthcare Institution "Departmental Clinical Hospital on Kemerovo Station of Public Corporation "Russian Railroad", Kemerovo, Russian Federation
  - Krasnodar regional hospital #1 n.a. Prof. Ochapovskiy S.V., Krasnodar, Russian Federation
  - Moscow State Healthcare Institution, City Clinical Hospital #15, Moscow, Russian Federation
  - First Moscow State Medical University, Moscow, Russian Federation
  - City Polyclinic # 109, Saint Petersburg, Russian Federation
  - City Hospital #38 named after Semashko N.A., Saint Petersburg, Russian Federation
  - Almazov Federal Heart, Blood And Endocrinology Centre, Saint Petersburg, Russian Federation
  - St. Petersburg State Health Care, Institution Pokrovskaya City Hospital, Saint Petersburg, Russian Federation
  - Tyumen Cardiology Center, Tyumen, Russian Federation
  - City Hospital #4, Vladimir, Russian Federation
  - Clinical Hospital n.a. N.V. Solovyov, Yaroslavl, Russian Federation
  - Ural Medical Academy, Yekaterinburg, Russian Federation
  - State Budgetary Healthcare Institution "State Novosibirsk Regional Clinical Hospital", Novosibirsk, Russia
  - Regional Cardiology Center, Volgograd, Russia
  - Smolensk State Medical Academy Of Roszdrav, Smolensk, Smoleskaya Oblast
  - Federal State Budgetary Institution Research Institution Of Cardiology Of Sibirsky, Tomsk, Tomskaya Obl.
- Ukraine (16):
  - Ivano-Frankivsk Regional Clinical Cardiology Dispensary, department of anesthesiology with intensive care unit, Ivano-Frankivsk, Ukraine
  - L.T. Malaya Therapy Institute of National Academy of Medical Sciences of Ukraine, Head of Cardiopulmonology Department Government Institution, Kharkiv, Ukraine
  - L.T. Malaya Therapy Institute of National Academy of Medical Sciences of Ukraine, Kharkiv, Ukraine
  - Institute Of Gerontology, Department Of Clinical Physiology And Pathology Of Internal Organs, Kiev, Ukraine
  - Kyiv Oleksandrivska Clinical Hospital, Kiev, Ukraine
  - Municipal Clinical Hospital #1, Kiev, Ukraine
  - National medical university named after O.O.Bogomolets, Kiev, Ukraine
  - Lviv Regional State Clinical Threatment-and-Diagnostic Cardiology Center, Lviv, Ukraine
  - Department of Family Medicine and General Practice of Odessa National Medical University, Odesa, Ukraine
  - City Clinical Hospital No. 3, Odesa, Ukraine
  - Odessa regional cardiological dispensary, Odesa, Ukraine
  - District Clinical Hospital Of Station "Uzhgorod", Dgto "Lviv Railway Station" Therapeutic Department, Uzhhorod, Ukraine
  - City Clinical Hospital # 1, Vinnitsa, Ukraine
  - Vinnytsya Regional Specialized Center for Radiation Protection of People, Vinnytsia, Ukraine
  - Regional medical center of cardiovascular diseases, Zaporizhzhya, Zaporizhzhia Oblast
  - Department of internal diseases #2, Zaporizhzhya, Zaporizhzhia Oblast

REFERENCES:
- [Derived] Shi Y, Liu D, Yuan J, Yan L, Zhan Z, Pan D, Lin L, Mu B. Compound Danshen Dripping Pills Prevented Leptin Deficiency-Induced Hepatic ER Stress, Stimulated Autophagy, and Improved Insulin Resistance of ob/ob Mice. Evid Based Complement Alternat Med. 2020 Jul 3;2020:5368657. doi: 10.1155/2020/5368657. eCollection 2020. PMID 32714408
- See also: manufacture and sponsor — http://www.tasly.com